CLINICAL TRIAL: NCT00695903
Title: A Phase 2 Multicenter, Randomized, Double-blinded, Study to Describe the Safety, Efficacy, and Pharmacokinetics of Daptomycin 10 mg/kg/Day and Vancomycin for the Treatment of Methicillin-resistant Staphylococcus Aureus Bacteremia
Brief Title: Phase 2 Study of Safety, Efficacy, and Pharmacokinetics of Higher Doses of Daptomycin and Vancomycin in MRSA Bacteremia
Acronym: HDSAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to lack of enrollment
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3009-013; DAP-HDSAB-07-05 (Other: Cubist Study Number)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Endocarditis, Bacterial; Infective Endocarditis
Keywords: Gram-positive bacterial infections; Staph Aureus; Bacteremia; MRSA; Infective Endocarditis; Right-sided Infective endocarditis; SABIE; SAIE; RIE
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis; Gram-Positive Bacterial Infections; Staphylococcal Infections; Bacteremia | interventions — Daptomycin; Injections; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- daptomycin 10 mg/kg (Experimental): Daptomycin 10 mg/kg IV every 24 hours
  Interventions: Drug: daptomycin
- vancomycin high-dose (Experimental): Vancomycin 15 mg/kg IV, dosed to maintain trough serum concentrations of 15 to 20 μg/mL
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: daptomycin — daptomycin 10 mg/kg IV every 24 hours
  Other Names: Cubicin; daptomycin for injection
  Arms: daptomycin 10 mg/kg
Drug: vancomycin — Vancomycin 15 mg/kg IV, dosed to maintain trough serum concentrations of 15 to 20 μg/mL
  Other Names: vancocin
  Arms: vancomycin high-dose

SUMMARY:
The overall goals of this study are to compare the safety and efficacy of daptomycin monotherapy 10 mg/kg/day and vancomycin monotherapy dosed to achieve vancomycin trough levels of 15 to 20 μg/mL for the treatment of methicillin-resistant S. aureus bacteremia (MRSA), including right-sided infective endocarditis (RIE).

DETAILED DESCRIPTION:
Patients who meet all inclusion criteria and exhibit none of the exclusion criterial will be randomized to one of two treatment arms:

1. daptomycin Intravenously (IV) 10 mg/kg every 24 hours
2. vancomycin IV dosed to maintain trough levels of 15 to 20 μg/mL.

The suggested duration of therapy with daptomycin or vancomycin will be 28 days (or up to 42 days if clinically indicated). Dose adjustments for both drugs will be made by an unblinded pharmacist at each site. To minimize the duration with which patients are treated with antibacterial agents effective against S. aureus prior to enrollment, patients with suspected MRSA bacteremia will be enrolled pending definitive culture results. Suspected MRSA bacteremia will be defined clinically or as initial blood cultures that grow Gram-positive cocci and that were obtained from a patient at increased risk for methicillin-resistant S. aureus infections. However, only patients with confirmed MRSA bacteremia or right-sided infective endocarditis will remain in the study and be evaluated for efficacy. During treatment, regular assessments will be performed. An End-of Therapy (EOT) will be performed 1-3 days after stopping therapy or upon Early Termination (ET). All patients will have a post therapy visit for Test of Cure (TOC) performed 35-49 days following last dose of study drug.

ELIGIBILITY:
INCLUSION CRITERIA:

* Written informed consent has been obtained;
* ≥18 years of age;
* Suspected MRSA bacteremia determined by clinical judgment or 2 sets of positive blood cultures;
* Increased risk for an MRSA infection

EXCLUSION CRITERIA:

* Received >48 hours of vancomycin therapy in the 7 days prior to enrollment;
* Received any systemic antibacterial agents potentially effective against MRSA in the 7 days prior to enrollment;
* Anticipated requirement of antibiotics potentially effective against MRSA;
* High likelihood of left-sided infective endocarditis (LIE);
* Known/suspected polymicrobial bacteremia or infection including Gram-negative infections;
* Known pneumonia, osteomyelitis, or meningitis;
* Intravascular foreign material unless material intended removed within 3 days;
* Prosthetic heart valve;
* Cardiac decompensation, valve damage, or both such that high likelihood of valve replacement surgery within first 3 days of study drug treatment;
* Moribund clinical condition such that death likely within first 3 days of study drug treatment;
* Shock or hypotension or oliguria unresponsive to fluids after 4 hours;
* Received investigational drug within 30 days of study entry
* Received statins or other therapy with associated with rhabdomyolysis within 2 days of study entry;
* History of significant allergy or intolerance to vancomycin or daptomycin
* Infecting pathogen with confirmed reduced susceptibility to vancomycin;
* Infecting pathogen with confirmed reduced susceptibility to daptomycin
* Creatinine clearance <30 mL/min (Cockcroft-Gault equation actual body weight)
* Serum creatine phosphokinase (CPK) ≥500 U/L
* Alanine transaminase (ALT) or aspartate aminotransferase (AST) >5 X ULN;
* Total bilirubin ≥3.0 mg/dL;
* Severe neutropenia or expected development severe neutropenia during study;
* Known or suspected HIV infection with a CD4+ T-cell count <200/μL;
* Unlikely to comply with study procedures or return for evaluations;
* Body Mass Index (BMI) ≥40 kg/m2;
* Pregnant or nursing;
* Female of childbearing potential not willing to practice barrier methods of birth control.

CONTINUATION CRITERIA:

* Fulfills A or B or both: A) Confirmed complicated MRSA bacteremia B) Possible or definite RIE caused by MRSA according to modified Duke criteria;
* Infecting S. aureus strain susceptible to vancomycin;
* Infecting S. aureus strain susceptible to daptomycin;
* Appropriate treatment of any foci of infection within first 3 days of study;
* Removal of any intravascular foreign material not allowed per inclusion criteria within first 3 days of study;
* Removal of any percutaneous or implanted catheters not allowed per inclusion criteria within first 3 days of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09-17 (Actual); Primary Completion 2010-08-24 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pertel, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (2):
- United States (2):
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin 10 mg/kg: Daptomycin 10 mg/kg Intravenously (IV) every 24 hours
Period: Had End of Therapy (EOT) Assessment
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Started | 19 | 19
Met Continuation Criteria | 9 | 6
Completed | 7 | 4
Not Completed | 12 | 15
Not completed — Randomized not treated | 0 | 2
Not completed — No confirmed MRSA | 9 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 2
Period: Had Test of Cure (TOC) Assessment
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Started | 7 | 4
Completed | 5 | 3
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Categorical [Count of Participants; unit: Participants] — Safety Population. Two patients in the high-dose vancomycin arm were randomized but not treated and therefore not included in the safety population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 16 | 15 | 31
    >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population. Two patients in the high-dose vancomycin arm were randomized but not treated and therefore not included in the safety population.
  Participants
    Female | 6 | 4 | 10
    Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Creatine Phosphokinase (CPK) Elevations
Description: Number of participants with treatment-emergent CPK elevations ≥5 x upper limit of normal (≥1,000 U/L) by the EOT visit.
Time Frame: On therapy and up to 3 days post-therapy (treatment duration ranged from 2 to 43 days)
Population: All subjects who received at least one dose of study medication (Safety Population). Two patients in the high-dose vancomycin arm were randomized but not treated and therefore not included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Number analyzed (Participants) | 19 | 17
Participants | 2 [2.9 to 31.4] | 0

2. Secondary Outcome: Number of Participants With Treatment Cure at End of Therapy (EOT) Visit
Description: Investigator's assessment of treatment cure. Treatment Cure includes successful outcomes of both clinical and microbiological assessments. Clinical cure is defined by clinical improvement of symptoms and signs associated with the underlying infection such that no further anti-infective therapy is required. Microbiological Success is defined by the eradication or presumed eradication of baseline infecting methicillin-resistant S. aureus pathogen and no superinfecting pathogen(s) (Gram-positive) or metastatic methicillin-resistant S. aureus pathogens were isolated post therapy.
Time Frame: End of Therapy (median day 12 and 6.5 in daptomycin and vancomycin modified intent-to treat population, respectively)
Population: Patients who met the continuation criteria (modified intent-to-treat) and had a EOT assessment of clinical outcome.
Measure: Number; unit: participants
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Number analyzed (Participants) | 7 | 4
participants | 6 [48.7 to 97.4] | 3 [30.1 to 95.4]

3. Primary Outcome: Number of Participants With Elevated Serum Creatinine
Description: Number of participants with treatment-emergent serum creatinine increases ≥0.5 mg/dL (for patients with a baseline value ≤3.0 mg/dL) or ≥1.0 mg/dL (for patients with a baseline value >3.0 mg/dL) by the EOT visit.
Time Frame: On therapy and up to 3 days post-therapy (treatment duration ranged from 2 to 43 days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Number analyzed (Participants) | 19 | 17
participants | 0 [NA to NA] | 4 [9.6 to 47.3]

4. Secondary Outcome: Number of Participants With Treatment Cure at Test of Cure (TOC)/Safety Visit
Description: Investigator's assessment of clinical response. Treatment Cure includes successful outcomes of both clinical and microbiological assessments. Clinical cure is defined by clinical improvement of symptoms and signs associated with the underlying infection such that no further anti-infective therapy is required. Microbiological Success is defined by the eradication or presumed eradication of baseline infecting methicillin-resistant S. aureus pathogen and no superinfecting pathogen(s) (Gram-positive) or metastatic methicillin-resistant S. aureus pathogens were isolated post therapy.
Time Frame: Test of Cure (TOC) Visit (35 to 49 days post-therapy, approximately week 8)
Population: Subset of modified intent-to-treat population who completed TOC/Safety visit
Measure: Number; unit: participants
Arm/Group | Daptomycin 10 mg/kg | Vancomycin High-dose
Number analyzed (Participants) | 5 | 3
participants | 5 [56.6 to 100.0] | 3 [43.9 to 100.0]

ADVERSE EVENTS:
Time Frame: Safety assessments were performed throughout the study (an average of 8 weeks). Safety assessments were conducted at the EOT/Early Termination visit (on the day of or within 3 days after therapy was stopped) and TOC visit (35 to 49 days post-therapy).
Description: On therapy safety assessments included maximum daily temperature, vital signs, physical examination and clinical laboratory tests. Investigators were required to report lab abnormalities (e.g. CPK, serum creatinine) as adverse events only when he/she considered the abnormality clinically significant.
Groups:
- Daptomycin: Daptomycin 10 mg/kg i.v.q24hr
- Vancomycin: Vancomycin 15 mg/kg i.v., dosed to maintain trough serum concentrations of 15 to 20 ug/mL
Arm/Group | Daptomycin | Vancomycin
Serious Adverse Events (participants affected / at risk) | 3/19 | 4/17
Other Adverse Events (participants affected / at risk) | 6/19 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=19) | Vancomycin (N=17)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin (N=19) | Vancomycin (N=17)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter related complication (General disorders) | 0 (0) | 1 (1)
Catheter site discharge (General disorders) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (2) | 0 (0)
Catheter site oedema (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 1 (3) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Because the study was terminated early due to lack of enrollment, there were not sufficient patients to provide meaningful analysis for the following secondary outcomes: persistent/recurrent bacteremia and time to defervescence/clearance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If first publication not published within 1 year of study conclusion or termination, Investigator has right to publish and disclose the data. Prior to any submission for publication, presentation, or communication of results or information arising from the study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.